CLINICAL TRIAL: NCT05104203
Title: Perioperative Analgesia Efectivity of Thoracolumbar Interfascial Plane Block Compared Modified Thoracolumbar Interfascial Plane Block in Posterior Lumbal Decompression and Stabilization: Research in Intraoperative Hemodynamic and qNox and Total Morfin Comsumption and Postoperative IL-6 Concentration
Brief Title: TLIP Block Versus Modified TLIP Block for Posterior Decompression and Stabilization Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Doctor, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes111
Record Dates: First submitted 2021-07-21; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Analgesia; Surgical Procedure, Unspecified
Keywords: Erector Spinae Plane Block; opioid consumption; numerical rating scale; Interleukin 10; Interleukin 6; Thoracolumbal Interfascial Plane Block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracolumbar Interfascial Plane block (Active Comparator): Patient will receive Thoracolumbar Interfascial Plane block
  Interventions: Procedure: Thoracolumbar Interfascial Plane block; Procedure: Modified Thorcolumbar Interfascial Plane block
- Modified Thoracolumbar Interfascial Plane block (Experimental): Patient will receive modified Thoracolumbar Interfascial Plane Block
  Interventions: Procedure: Thoracolumbar Interfascial Plane block; Procedure: Modified Thorcolumbar Interfascial Plane block

INTERVENTIONS:
Procedure: Thoracolumbar Interfascial Plane block — Interfascial block done by injection between m. multifidus and m. longissimus
Procedure: Modified Thorcolumbar Interfascial Plane block — Injection of local anesthetics between m. longissimus and m. illiocostalis

SUMMARY:
This study aimed to compare the analgesia effectivity of TLIP and modified TLIP block in Posterior Lumbar Decompression and Stabilization Surgery Perioperatively.

DETAILED DESCRIPTION:
This study aimed to compare the analgesia effectivity of TLIP and modified TLIP block in Posterior Lumbar Decompression and Stabilization Surgery. Intraoperatively, total fentanyl consumption, hemodynamic, and mean qNox Score was recorded. And Postoperatively, the patient was given the PCA, and total morphine consumption was assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergo thoracolumbar Decompression and Stabilization Surgery
2. Age between 18-65 years old
3. BMI >18,5 kg.m2, and BMI< 30 kg/m2
4. ASA 1-3
5. No contraindications for the patients to do the Block, and the patients agree and signed the informed consent before the procedure was done

Exclusion Criteria:

1. Obese patient, with BMI>30 kg.m2
2. Alergic to local anesthetics
3. Underweight patient with BMI <18,5 kg/m2"

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Hemodynamic | approximately 15 minutes within surgery
  Stability of Hemodynamics that needs the fentanyl addition

SECONDARY OUTCOMES:
qNox Score | before induction of anesthesia, 15, 30, 45 minutes after the block was done.
  qNox score were taken before induction of anesthesia, 15, 30 and 45 minutes after the block done. the mean of 15,30 and 45 minutes qNox score was assesed

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided